CLINICAL TRIAL: NCT06504511
Title: SCN1A Horizons A Natural History Study of SCN1A-related Epilepsies in the United Kingdom
Status: Recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN20NE522P; 295069 (Other: IRAS); 316675 (Other: IRAS)
Record Dates: First submitted 2024-06-04; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: SCN1A; Dravet Syndrome; Epilepsy
Keywords: Epilepsy; SCN1A; Natural History; Developmental Outcome
MeSH Terms: conditions — Epilepsies, Myoclonic; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2x 4ml EDTA blood sample at baseline visit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aims of this prospective natural history study are to define the seizure, neuro-developmental, and behavioural characteristics of SCN1A-related epilepsies/Dravet syndrome in children and adults longitudinally over a period of three years. In addition, this study will compare missense and truncating genotypes in terms of i) rates of change of countable convulsive seizures per month and ii) neurodevelopmental outcome and trajectories.

DETAILED DESCRIPTION:
Our aim is to define the seizure, neurodevelopmental, and behavioural characteristics of SCN1A-related epilepsies/Dravet syndrome in children and adults longitudinally over a period of three years. In addition, this study will compare missense and truncating genotypes in terms of i) rates of change of countable convulsive seizures per month and ii) rate of change in neurodevelopmental outcomes over time. The investigators will therefore prospectively study the natural history of SCN1A-related epilepsies and Dravet syndrome in the UK. In order to explore established and novel treatments, including new medications, it is important to not only document seizure frequency but also behaviour, learning and motor function. Treatment interventions are key to prevent the neurodevelopmental comorbidities of Dravet syndrome; as such sensitive measures of disease progression and a clear prospective description of the natural history of the disease across the lifespan is required to know whether therapies are transformative.

Although the decline in neurodevelopmental profile and motor function in patients with SCN1A-related epilepsies/Dravet syndrome have been described, no large scale long-term, prospective studies of cognition and motor function have been conducted in SCN1A-related epilepsies/Dravet syndrome with established measures.

The SCN1A/Dravet syndrome natural history study will provide a platform to systematically collect longitudinal validated outcome measures for SCN1A variant-carrying patients across the UK. The study will prospectively assess changes in cognition, behaviour, and quality of life, as well as other co-morbidities.

A number of important questions relating to the natural history of SCN1A-related epilepsies/Dravet syndrome over the lifespan remain unanswered:

* It is not understood the precise neurodevelopmental profile and decline of individuals with SCN1A-related epilepsies over time and which factors might modify this?
* There are no reliable biomarkers that can inform disease severity or treatment planning
* What impact does the underlying genotype have on the neurodevelopmental outcome?
* Do clinical features such as the occurrence of repeated episodes of status epilepticus and/or contraindicated medication use worsen the neurodevelopmental outcome?
* What is the seizure burden across different ages and does treatment response change over the lifespan?
* There is a lack of understanding of the comorbidity profile that individuals with SCN1A-related epilepsies experience over the lifespan
* More information is required on the socio-economic impact SCN1A-related epilepsies have on affected individuals, families and society

ELIGIBILITY:
Patients meeting the following inclusion criteria will be considered eligible for this study:

1. Patient and/or legally authorised representative must be willing and able to give informed consent/assent for participation in the study.
2. Patient and parent/caregiver are willing and able (in the Investigator's opinion) to comply with all study requirements (including ability and willingness to comply with virtual visits).
3. Participant has a confirmed pathogenic (class 5) or likely pathogenic (class 4. SCN1A variant, as demonstrated by genetic testing.

Exclusion criteria:

Patient has any other significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or may affect the patient's ability to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 400 participants with a minimum of 2 years of follow-up are planned to be enrolled. Recruitment will be stratified according to the following age distribution:
  * 300 patients in the Comprehensive study arm (clinical and face-to-face neurodevelopmental assessments)
    * Approximately 60 participants aged 6 to 35 months
    * Approximately 80 participants aged 3 to 6 years inclusive
    * Approximately 100 participants aged 7 to 16 years inclusive
    * Approximately 60 participants aged 17 years and older
  * 100 patients in the Basic study arm (clinical and non-face-to-face neurodevelopmental assessments), in case the age specific quota in the Comprehensive study arm has been filled.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Countable convulsive seizures per month | Up to 3 year follow up
  A 4-week seizure diary will be completed by caregivers or participants (where they have capacity to do so) every 6 months.
Bayley Scales of Infant and Toddler Development 4th UK Edition (Bayley-4) | Administration will occur 6-monthly for patients <7 years old and 12-monthly for patients 7 years and older. There is a planned 2-3 year follow up.
  Patients in the comprehensive arm who are <30 months of age will be administered the Bayley-4. Participants older than 30 months old may be administered the Bayely-4 if they are unable to access age-appropriate assessment. Standard scores range from 45-155 on each domain (cognitive, language & motor). Growth Scale Values range from 428-559. Higher scores are indicative of higher developmental functioning.
Wechsler Preschool and Primary Scale of Development 4th UK Edition (WPPSI-IV) | Administration will occur 6-monthly for patients <7 years old and 12-monthly for patients 7 years and older. There is a planned 2-3 year follow up.
  Patients in the comprehensive arm who are ≥2 years 5 months and ≤6 years of age will be administered the WPPSI-IV at Baseline. If the patient is unable to access the WPPSI-IV, they will be administered the Bayley-4 in addition to the WPPSI-IV at Baseline. Composite score for each domain ranges from 45-155. Composite full scale score ranges from 40-160. Higher scores are indicative of higher developmental functioning.
Wechsler Intelligence Scale for Children 5th UK Edition (WISC-V) | Administration will occur 6-monthly for patients <7 years old and 12-monthly for patients 7 years and older. There is a planned 2-3 year follow up.
  Patients in the comprehensive arm aged 6 years to 16 years will be administered the WISC-V at baseline. If the patient is unable to access the WISC-V they will be administered the WPPSI-IV in addition to the WISC-V at Baseline. Participants will drop down to the Bayley-4 if they are unable to access the WPPSI-IV. Administration will occur 6-monthly for patients <7 years old and 12-monthly for patients 7 years and older. Composite score for each domain ranges from 45-155. Composite full scale score ranges from 40-160. Higher scores are indicative of higher developmental functioning.
Wechsler Adult Intelligence Scale 4th UK Edition (WAIS-IV) | Administration will occur 12-monthly. There is a planned 2-3 year follow up.
  Patients in the comprehensive arm aged 16 years and older will be administered the WAIS-IV, 12-monthly. Composite score for each domain ranges from 50-150. Composite full scale score ranges from 40-160. Higher scores are indicative of higher developmental functioning.
Vineland Adaptive Behaviour Scales - Third Edition | Participants age <7 will have a Vineland assessment completed every 6 months, participants age 7 years and older will have a Vineland assessment completed every 12 months.
  All patients in the comprehensive and basic arm will be administered the Vineland Adaptive Behaviour Scales - Third Edition, which will be completed by the caregiver. Raw scores range from 0-116. Standard scores range from 20-140. Growth Scale Values range from 10-197. Higher scores are indicative of higher developmental functioning.

SECONDARY OUTCOMES:
Occurrence and frequency of status epilepticus | Up to 3 year follow up
  Information obtained during 6-monthly standard of care clinical visit with Consultant Paediatric Neurologist for all patients.
Grantham Score | Baseline
  A measure of physiochemical difference between amino acids. The score can range from 5-215, with a higher score indicative of more radical change in amino acid properties.
Combined Annotation Dependent Depletion (CADD) score | Baseline
  Score of the deleteriousness of single nucleotide variants and insertion/deletion variants in the human genome. The score can range from 1-99, with higher values indicating more deleterious cases.
Rare Exam Variant Ensemble Learner (REVEL) score | Baseline
  Predicts the pathogenicity of missense variants. The score can range from 0-1, with higher scores indicating a higher likelihood of the variant being disease-causing.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Brunklaus, MD PhD, Principal Investigator — NHS Greater Glasgow & Clyde
Locations (1):
- Royal Hospital for Children, Glasgow, United Kingdom